CLINICAL TRIAL: NCT03039634
Title: A Multicenter, Double-blind, Nontreatment, Long-term, Follow-up Study of Subjects Who Completed Clinical Studies 755.1100_FA, 810.1100_FA, or 1064.1100_FA of a Topical Silver Particle Solution Followed by Laser for the Treatment of Facial Acne Vulgaris
Brief Title: Long-term Follow-up Study of Subjects Who Completed Clinical Studies 755.1100_FA, 810.1100_FA, or 1064.1100_FA
Status: Completed | Type: Observational
Sponsor: Sienna Labs (Industry)
Responsible Party: Sponsor
Other Study IDs: SL-2016-01_FA
Record Dates: First submitted 2017-01-25; First posted 2017-02-01 (Estimated); Last update posted 2019-03-04 (Actual); Status verified 2018-05

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study evaluates the safety, effectiveness, and maintenance of effect of a novel topical silver particle solution (Sienna 755.1100, 810.1100, or 1064.1100) used in conjunction with a laser for the treatment of Acne Vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Subject has participated in study 755.1100_FA, 810.1100_FA, or 1064.1100_FA and fulfilled that study's exit criteria (ie, completion of the final visit [visit 7] of that study).
* Subject has followed predecessor study restrictions prior to study entry.
* Subject is able to provide informed consent and Health Insurance Portability and Accountability Act (HIPAA); minors will in addition have parent or legal guardian provide consent.
* Subject is willing to comply with the schedule, procedures, and restrictions of the study.

Exclusion Criteria:

* Subjects who have had any treatments or conditions (eg, pregnancy or metabolic disease) that may affect assessment of the safety or efficacy since enrollment in the predecessor study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 165 subjects will be considered for entry into the study. Subjects completing a predecessor facial acne study (755.1100_FA, 810.1100_FA, or 1064.1100_FA) who meet all study inclusion/exclusion criteria will be offered study participation. There will be no treatments administered in this study.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2016-08; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Change in Total lesion count by blinded investigator | 18 weeks post final treatment
  Maintenance of effect by comparing lesion counts conducted at the exit visit of the predecessor study (ie, 12 weeks post-final treatment) and visit 2 of this study (ie, 18 weeks post-final treatment).
Change in Total lesion count by blinded investigator | 24 weeks post final treatment
  Maintenance of effect by comparing lesion counts conducted at the exit visit of the predecessor study (ie, 12 weeks post-final treatment) and visit 3 of this study (ie, 24 weeks post-final treatment).
Safety as assessed by number of adverse events | up to 24 weeks post final treatment
  Adverse events will be monitored throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Paul Lizzul, MD, Study Director — Sienna Biopharmaceuticals
Locations (16):
- United States (16):
  - Scottsdale, Arizona
  - Santa Monica, California
  - Coral Gables, Florida
  - Miami, Florida
  - Hunt Valley, Maryland
  - Beverly, Massachusetts
  - St Louis, Missouri
  - Hackensack, New Jersey
  - Charlotte, North Carolina
  - Yardley, Pennsylvania
  - Charleston, South Carolina
  - Houston, Texas
  - Pflugerville, Texas
  - San Antonio, Texas
  - Jordan, Utah
  - Spokane, Washington

IPD SHARING:
Plan to Share IPD: No